CLINICAL TRIAL: NCT00399204
Title: A Randomised Pilot Study to Compare the Effect of Pioglitazone and Metformin on Cardiovascular Morbidity and Mortality in Patients With Type 2 Diabetes
Brief Title: Comparison of Cardiovascular Outcomes of Pioglitazone and Metformin in Type 2 Diabetes Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Council of Scientific and Industrial Research, India (Other Government)
Responsible Party: Principal Investigator, SHotra, professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pharma6/701
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- Control (Active Comparator): Metformin
  Interventions: Drug: Pioglitazone vs Metformin
- Experimental (Experimental): Pioglitazone
  Interventions: Drug: Pioglitazone vs Metformin

INTERVENTIONS:
Drug: Pioglitazone vs Metformin

SUMMARY:
The study aims to see if there is any significant difference in the cardiovascular outcomes in type 2 diabetes patients who are treated with pioglitazone or Metformin

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed (less than six months since diagnosis and not controlled on dietary modifications) type 2 diabetic patients of both sexes aged 25-60 years.
2. Ready to give written informed consent

Exclusion Criteria:

1. Presence of ketonuria
2. Severe concurrent, infection or illness
3. History of hypersensitivity to any study drug
4. Impaired renal function
5. Pulmonary insufficiency with hypoxemia
6. Severe hepatic disease
7. Congestive heart failure
8. History of myocardial infarction or angina(stable/unstable)
9. History of alcohol or drug abuse
10. Pregnant or lactating women -

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01 (Estimated); Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Promila Pandhi, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh; Nusrat Shafiq, MD,DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Anil Bhansali, MD,DM, Study Director — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, India